CLINICAL TRIAL: NCT05478538
Title: Observational Lung Trial to Collect Tissue to Train and Validate a Live Tumor Diagnostic Platform (CYBRID-01)
Brief Title: Observational Lung Trial to Collect Tissue to Train and Validate a Live Tumor Diagnostic Platform
Acronym: CYBRID-01
Status: Recruiting | Type: Observational
Sponsor: Elephas (Industry)
Responsible Party: Sponsor
Other Study IDs: ELEP-2022-CYBRID-01
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: NSCLC (Non-small Cell Lung Cancer); Metastatic NSCLC - Non-Small Cell Lung Cancer
Keywords: Metastatic NSCLC; NSCLC; Non Small Cell Lung Cancer; Core needle biopsy; Live tumor fragments; Immunotherapy; Immunotherapy prediction; 3D culture; Ex vivo platform; Immune checkpoint inhibitors; Forceps biopsy; Punch biopsy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Biopsy, Needle; Surgical Instruments

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tissue sampling using core needle, forceps, or punch biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage IV or metastatic Non Small Cell Lung Cancer (NSCLC): Subjects suspected of or diagnosed with Stage IV NSCLC and meet one of the following criteria:
  1. Subjects who are undiagnosed, have undergone imaging and are suspected to have Stage IV lung cancer.
  2. Subjects with a Stage I, II, or III diagnosis of NSCLC, who are being re-biopsied after imaging-confirmed progression to metastatic disease
  3. Subjects who have a confirmed diagnosis of NSCLC, and have undergone a SOC biopsy procedure and will undergo a separate procedure for the purposes of this study.
  4. Subjects who have a previous Stage IV/metastatic NSCLC diagnosis and have already received first line treatment.
  Interventions: Procedure: Core Needle, Forceps, or Punch Biopsy

INTERVENTIONS:
Procedure: Core Needle, Forceps, or Punch Biopsy — Subjects must be clinically able, at investigator discretion, to undergo additional core needle, forceps, or punch biopsy during their biopsy. These additional biopsies may either be collected from the primary tumor or a metastatic site amenable to additional passes (e.g., liver or lymph nodes) per the clinician.

SUMMARY:
The primary objective of this study is to determine the ex-vivo prognostic accuracy of the Cybrid live tumor diagnostic platform using in-vivo RECIST 1.1 as the reference method.

DETAILED DESCRIPTION:
Cancer is a leading cause of death and despite many new drugs, a major diagnostic challenge remains knowing which drug will work best for a patient. A new class of drugs called immune checkpoint inhibitors (ICIs) have revolutionized cancer treatment. However, current diagnostic methods (e.g. PDL1, MSI and TMB) do not accurately predict which patients will respond.

Elephas is developing a diagnostic platform using small 3D Live Tumor Fragments (LTFs) from participants for accurate prediction of drug response with a focus on ICIs such as Pembrolizumab (Keytruda). These LTFs contain both tumor cells and infiltrating immune cells, which are critical in determining response to ICIs and other immunotherapies.

In this observational clinical trial, 200 Non-Small Cell Lung Cancer (NSCLC) participants will be recruited and their actual clinical response to ICIs (using RECIST 1.1) will be compared to the platform's predictive Artificial Intelligence (AI) score that is based on RNA, clinical data, and 3D microscopy images. The sensitivity and specificity of the platform's score will be determined and compared to current diagnostic methods for ICIs like PDL1, MSI, and TMB.

ELIGIBILITY:
Subject Inclusion Criteria

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. Subjects suspected of or diagnosed with Stage IV/metastatic NSCLC and meet one of the following criteria:

   1. Subjects who are undiagnosed, have undergone imaging and are suspected to have Stage IV lung cancer.
   2. Subjects with a previous Stage I, II, or III diagnosis of NSCLC, who are being re-biopsied due to suspected progression to metastatic disease.
   3. Subjects who have a newly confirmed diagnosis of Stage IV NSCLC, have undergone a SOC biopsy procedure and will undergo a separate procedure for the purposes of this study prior to starting first line treatment.
   4. Subjects who have a previous Stage IV/metastatic NSCLC diagnosis and have already received first line treatment.
4. Subjects must be clinically able, at investigator discretion, to undergo additional CNB or forceps biopsy passes during their biopsy. These additional biopsies may either be collected from the primary tumor or a metastatic site amenable to additional passes (e.g., liver or lymph nodes) per the clinician.
5. Subjects who are newly diagnosed or have suspected cancer must be treatment-naïve at the time of biopsy. All other subjects should have the biopsy performed before starting their next line of treatment.

Subject Exclusion Criteria

1. Any patient for whom an extra biopsy might pose a clinical risk based on the discretion of the clinician.
2. Any mental impairment that would render the patient unable to understand his/her participation in the study would disqualify the patient from consenting and participating.
3. Subjects with an auto-immune disease that would render them ineligible for immune- oncology treatment.
4. Immunocompromised subjects, and subjects known to be HIV positive and currently receiving antiretroviral therapy. NOTE: Patients known to be HIV positive, but without clinician evidence of an immunocompromised state, are eligible for this trial.
5. Subjects who are enrolled or plan to be enrolled in a blinded oncology treatment trial are not eligible.
6. Subjects who are pregnant are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of or diagnosed with metastatic non-small cell lung cancer (NSCLC).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Cybrid Score for Predicting In-Vivo Clinical Response to Immune Checkpoint Inhibitors | 3 years
  The ex-vivo prognostic accuracy of the Cybrid live tumor diagnostic platform will be determined using in-vivo RECIST 1.1 as the reference method.

SECONDARY OUTCOMES:
Determine the Area Under the Receiver Operating Characteristic Curve (AUC) of Cybrid Score and Compare to the AUCs of Current FDA Approved Predictive Biomarkers PD-L1 and Tumor Mutation Burden (TMB) | 3 years
  The AUC of Cybrid Score will be established with a clinically meaningful confidence interval and compared to the AUCs of established FDA approved biomarkers for predicting clinical response to ICIs.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Hausheer, MD, FACP, Study Director — Elephas
Locations (7):
- United States (7):
  - UCLA Medical Center, Los Angeles, California
  - James M Stockman Cancer Institute, Frederick, Maryland
  - New York Cancer & Blood Specialists, Shirley, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - JPS Health Network, Fort Worth, Texas
  - Baylor Scott & White Research Institute, Temple, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Chen S, Zhang Z, Zheng X, Tao H, Zhang S, Ma J, Liu Z, Wang J, Qian Y, Cui P, Huang D, Huang Z, Wu Z, Hu Y. Response Efficacy of PD-1 and PD-L1 Inhibitors in Clinical Trials: A Systematic Review and Meta-Analysis. Front Oncol. 2021 Apr 16;11:562315. doi: 10.3389/fonc.2021.562315. eCollection 2021. PMID 33937012
- [Background] Cherukuri AR, Lubner MG, Zea R, Hinshaw JL, Lubner SJ, Matkowskyj KA, Foltz ML, Pickhardt PJ. Tissue sampling in the era of precision medicine: comparison of percutaneous biopsies performed for clinical trials or tumor genomics versus routine clinical care. Abdom Radiol (NY). 2019 Jun;44(6):2074-2080. doi: 10.1007/s00261-018-1702-1. PMID 30032384
- [Background] Basumallik N, Agarwal M. Small Cell Lung Cancer. 2023 Jul 10. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482458/ PMID 29494065
- [Derived] Ramasubramanian TS, Adstamongkonkul P, Scribano CM, Johnson C, Caenepeel S, Hrycyniak LCF, Vedder L, Dana N, Baltes C, Browning T, Chen YI, Dietz T, Flietner E, Kaplewski N, Kellner A, Korrer M, Liu C, Marhefke N, McDonnell P, Nasreen A, Pope V, Prasad A, Richardson J, Schneider S, Schultz M, Sood C, Sunil A, von Euw E, Wait E, Wargowski E, Advani P, Broome B, Bruckbauer A, Godwin A, Kokabi N, Martin R, Robaina M, Toia G, Routh J, Friedl A, Eliceiri K, Szulczewski M, Johnson S, Oliner J, Galon J, Capitini C, Mukhopadhyay D, Taube J, Braun D, Gierman HJ. A live tumor fragment platform to assess immunotherapy response in core needle biopsies while addressing challenges of tumor heterogeneity. bioRxiv [Preprint]. 2025 Jul 18:2025.07.18.663728. doi: 10.1101/2025.07.18.663728. PMID 40791544